CLINICAL TRIAL: NCT06313671
Title: Reliability of Plethysmographic Perfusion Index to Predict Fluid Responsiveness in Acute Circulatory Failure.
Brief Title: Plethysmographic Perfusion Index and Fluid Responsiveness
Acronym: PPI-FR
Status: Completed | Type: Observational
Sponsor: Avicenna Military Hospital (Other)
Responsible Party: Principal Investigator, Younes Aissaoui, MD, Professor of Anesthesiology and Intensive Care Medicine - Head of intensive care unit, Avicenna Military Hospital
Other Study IDs: Perfusion Index - FR study
Record Dates: First submitted 2024-01-07; First posted 2024-03-15 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Fluid Responsiveness
Keywords: acute circulatory failure; fluid responsiveness; perfusion index; left ventricular outflow velocity time-integral; echocardiography
MeSH Terms: conditions — Shock | interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Perfusion index — The perfusion index (PI) is derived from the plethysmography signal and represents the ratio of pulsatile to non-pulsatile light absorbance of the plethysmography signal.
  PPG signal.

SUMMARY:
The objective of this study is to assess the reliability of the perfusion index to predict fluid responsiveness in patients with acute circulatory failure in intensive care.

DETAILED DESCRIPTION:
In patients with acute circulatory failure, it is recommended to assess fluid responsiveness. Fluid responsiveness is defined by an increase in cardiac output of 10 to 15% after fluid loading. The assessment of fluid responsiveness usually needs cardiac output monitoring (or stroke volume). However, in limited resource settings or during the initial management of patients with acute circulatory failure, cardiac output measurement is usually unavailable. The perfusion index (PI) is derived from the plethysmographic signal of the pulse oximeter and represents the ratio between the ratio of pulsatile on non-pulsatile light absorbance of the plethysmography signal. The PI is influenced by vascular and stroke volume. The investigators hypothesized that the peripheral index could track the changes in cardiac output induced by fluid loading and therefore detect fluid responsiveness.

Adult patients with acute circulatory failure in whom physicians want to test the fluid responsiveness will be included. At baseline, the PI will be recorded. An initial echocardiography will be performed to measure the left ventricular outflow tract velocity time integral (a surrogate of stroke volume). A fluid loading with 500 ml of 0.9% Saline or Ringer Lactate will be performed. After fluid administration, the velocity time integral and the PI will be collected. Fluid-responsive patients are defined by a 15% increase in velocity time integral. The investigators will analyze the ability of the PI to detect fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 and older with acute circulatory failure (ACF).

Exclusion Criteria:

* Low echogenicity: the inability to perform echocardiographic measurements according to established recommendations.
* Absence of the plethysmographic signal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 and older with acute circulatory failure (ACF). ACF is defined by the presence of signs of tissue hypoperfusion: capillary refill time>5 seconds, mottling, oliguria <0.5 mL/kg/h for more than an hour), altered mental status), blood lactate >2 mmol/L or metabolic acidosis (pH <7.35 or base excess >-5). Arterial hypotension is not necessary for the diagnosis of ACF. It is defined by a systolic blood pressure (SBP) <90 mmHg, a mean arterial pressure (MAP) <65 mmHg, or a drop in SBP ≥40 mmHg. Shock is defined by the combination of ACF and arterial hypotension.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Reliability and accuracy of the perfusion index to discriminate fluid-responsiveness. | through study completion, an average of 9 months.
  Reliability and accuracy of the change in perfusion index to discriminate fluid-responsive patients. Fluid responsiveness is defined by an increase in the left ventricular outflow tract velocity time integral by 15% after fluid loading.

CONTACTS AND LOCATIONS:
Locations (1):
- Avicenna Military Hospital, Marrakesh, Marrakesh Tensift El Haouz, Morocco

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After study completion for 2 years
Access Criteria: University members Healthcare providers